CLINICAL TRIAL: NCT03655184
Title: An Observation Study on Neuropsychology and Serum Melatonin Level in Patients With Medication Overuse Headache
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-SR-239
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2018-08

CONDITIONS: Medication Overuse Headache
Keywords: melatonin; medication Overuse Headache; migraine; Neuropsychology
MeSH Terms: conditions — Headache Disorders, Secondary; Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples were stored at -70 ℃
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MOH group: Patients with medication overuse headache
- Episodic migraine group: Patients with episodic migraine
- Healthy group: No headache or other special medical history

SUMMARY:
Medication overuse headache (MOH) is a disabling and costly disorder which is characterized by chronic headache and overuse of different headache medications. Patients with MOH are more likely to coexist with affective disorders such as anxiety and depression, and are more likely to suffer from sleep disturbances than those with episodic headache.

Melatonin is a hormone secreted from the pineal gland. Melatonin is an antioxidant, antinociceptive, hypnotic, anticonvulsant, neuroprotective, anxiolytic, sedative and analgesic.

This observational study aims to investigate clinical characteristics of patients with MOH and to explore the relationship between the serum melatonin level and medication overuse headache. Researchers hope to provide a new idea for the clinical treatment of MOH: melatonin can be used as an adjuvant therapy for MOH in the future.

DETAILED DESCRIPTION:
30 patients with MOH，30 patients with episodic migraine and 30 age-matched healthy volunteers were recruited in the study. A series of neuropsychological test scale including Hospital Anxiety and Depression Scale (HADS), Pittsburgh sleep quality index (PSQI) and Leeds Dependence Questionnaire (LDQ) were evaluated among all the recruited. Blood samples were taken at 10 a.m. and centrifuged. The serum was separated and collected at -70 °C for the measurement of melatonin .

ELIGIBILITY:
Inclusion Criteria:

* Subject has medication overuse headache. Headache occurring on 15 or more days per month for more than 3 months. The number of medication days ≥10 days/month for triptans, ergotamine, opioids, combination analgesics, or multiple drug classes not individually overused; ≥15 days/ month for simple analgesic
* Subject has had 1-8 migraines per month over the previous 3 months
* Sign the informed consent

Exclusion Criteria:

* Subjects combine with other pain syndromes and long-term oral analgesics are needed
* History of bleeding disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients and inpatients in the First Affiliated Hospital of Nanjing Medical University
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-09-10 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum melatonin level | 30 minutes
  Blood samples taken for melatonin were centrifuged, and the serum content was separated and collected for analysis at -70 °C.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 15 minutes
  The subscore of HADS >7 is considered as possible anxiety or depression.
Pittsburgh sleep quality index (PSQI) | 15 minutes
  An overall score over 5 indicates poor sleep.
Leeds Dependence Questionnaire (LDQ) | 15 minutes
  The LDQ is a 10-item, self completion questionnaire designed to measure dependence upon a variety of substances.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Wan, professor, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Department of Neurology, the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tao H, Wan Q, Sun M, Cai K, Song Y, He M, Shen J. Involvement of Plasma Melatonin in Medication-Overuse Headache: A Cross-Sectional Study. Clin Neuropharmacol. 2024 Jan-Feb 01;47(1):12-16. doi: 10.1097/WNF.0000000000000573. Epub 2023 Oct 19. PMID 37852214